CLINICAL TRIAL: NCT06343272
Title: Effects of a Supplementation With a Mixture of Essential Amino Acids on Enhancing the Number of Circulating Lymphocytes and Improveing the Tolerance to Chemotherapy Treatment in Patients With Advanced Gastroinmtestinal Malignances the LEGO Trial
Brief Title: Lymphocyte Enhancement in Gastroenteric Oncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEGO
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Advanced Gastrointestinal Cancers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sperimental (Experimental)
  Interventions: Dietary Supplement: EAA supplementation
- Isocaloric placebo (Placebo Comparator)
  Interventions: Other: Isocaloric placebo

INTERVENTIONS:
Dietary Supplement: EAA supplementation — The experimental group will receive the mixture (Amino-Ther® PRO, Professional Dietetics, Milan) composed of (in mg): L-leucine 1200, l L-isine 900, L-threonine 700, L-isoleucine 600, L-valine 600, L-cystine 150, L histidine 150, L-phenylalanine 100, L-methionine 50, L-tryptophan 50, vitamin B6 0.85, vitamin B1 0.70, citric acid 409, acidomalic 102.5, succinic acid 102.5.
  1 sachet dissolved in 150 ml of water at 10.00 am +1 sachet at 4.00 pm daily for 60 days There are: proteins 0.00 g, carbohydrates 2.1 g, fats 0.00 g
  Arms: Sperimental
Other: Isocaloric placebo — The control group will take 25g of maltodextrins daily with the same methods as the treated group: 1 sachet dissolved in 150 ml of water at 10.00 am +1 sachet at 4.00 pm daily for 60 days
  Arms: Isocaloric placebo

SUMMARY:
LEGO is single center double-blind randomized trial aimed at testing the efficacy of an essential ammino acid (EAA) supplementation in improving the absolute count of peripheral lymphocytes and the tolerance to chemotherapy in patients with advanced gastrointestinal malignancies not candidates to immune check-point inhibitors containing regimens.

DETAILED DESCRIPTION:
The aim of the study is to verify that, in lymphopenic patients, AAE supplementation leads to an increase in lymphocytes circulating in the blood. In particular, at the end of treatment, in patients with lymphocytes < 29.7% of the total number of white blood cells, we want to observe the disappearance of lymphopenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of epithelial neoplasia of the gastrointestinal tract in advanced stage with indication for first-line chemotherapy for palliative purposes and with circulating lymphocytes < 29.7% of the number total white blood cells in the blood.
* ECOG PS ≤ 2
* start of first-line palliative chemotherapy agreement with AIOM guidelines.
* adequate nutritional counseling carried out before starting of the treatment
* willing to participate by providing written informed consent

Exclusion Criteria:

* age < 18 years
* current or indicated artificial nutrition
* gluten intolerance
* prediction of use of granulocyte growth factors
* confirmed diagnosis of COPD, chronic heart failure, insufficiency chronic kidney disease, chronic liver failure, collagen disease, diseases endocrine, insulin-dependent diabetes, malignancy in other locations. All these conditions are associated with documented alterations in the plasma profile of amino acids and potentially of subsets of circulating T lymphocytes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Exit from lymphopenia | 60 days
  Proportion of patients exceeding the lymphopenia threshold level of 29.7%.

SECONDARY OUTCOMES:
The change in the % of lymphocytes over time | 0, 30, 60, 90 days
  The change in the % of lymphocytes over time
The proportion of patients with G3-G5 toxicity | 60 days
  The proportion of patients with G3-G5 toxicity
The percentage of chemotherapy dose administered compared to that expected for the patients. | 60 days
  The percentage of chemotherapy dose administered compared to that expected for the patients.
plasma aminoacids composition chang during treatment | 60 days
  The proportion of patients experiencing a ≥10% reduction in lactate, acetoacetate and a >/= 10% increase in essential amino acids in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy